CLINICAL TRIAL: NCT07394049
Title: Cardiovascular Assesment Under Current Hormone Replacement Therapy in Menopause (CATCH-Menopause)
Brief Title: Impact of New Hormone Replacement Therapy After Menopause on Heart Health in Women
Acronym: CATCH-Menopaus
Status: Not yet recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: Catch-menopause
Record Dates: First submitted 2026-02-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hormone Replacement Therapy; Cardiovascular Diseases; Hormone Replacement Therapy, Post-Menopausal; Menopause
Keywords: hormone replacement therapy; cardiovascular disease; menopause
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — prospectively defined blood sampling protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post menopausal women with hormone replacement therapy: Postmenopausal women who have been in menopause and have taken any hormone replacement therapy (HRT).
- Post menopausal women without hormone replacement therapy (Control): Postmenopausal women who have been in menopause and have not taken any hormone replacement therapy (HRT) These participants serve as the control cohort to compare outcomes against those receiving HRT.

SUMMARY:
This prospective registry study investigates the impact of new hormone replacement therapy (HRT) delivery methods, such as creams, gels, and sprays, on cardiovascular risk in postmenopausal women. Menopause-related estrogen deficiency leads to metabolic and vascular changes that increase atherosclerosis and cardiovascular events. This study hypothesizes that new HRT forms may reduce cardiovascular risk in high-risk women."

DETAILED DESCRIPTION:
Detailed Description:

This prospective, longitudinal registry study will enroll peri- and postmenopausal women aged 45-75 years with cardiovascular disease, peripheral or cerebrovascular disease, a SCORE2 >5%, evidence of coronary artery disease progression, and who are receiving hormone replacement therapy (HRT). Age-matched postmenopausal women not receiving HRT will serve as controls.

Participants will be recruited from outpatient gynecology, cardiology and endocrinology clinics and followed for 10 years, with pseudonymized data collected on clinical events, cardiovascular and menopausal risk factors, lifestyle, lab values, and HRT details.

Blood samples will be collected during routine care with additional tubes for hormone and inflammatory marker analyses, and biobanking for up to 10 years. Follow-up visits will occur at 6 months and 1 year, with re-evaluation of clinical events, risk factors, menopausal symptoms, and HRT. Asymptomatic participants will not undergo additional testing.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75 years
* Score 2 > 5%
* Or existing coronary heart disease
* Or cAVK
* Or PAD

Exclusion Criteria:

* Age <45 years / > 75 years
* Existing cancer
* Language barrier, inability to provide informed consent
* GFR <30 ml/min or dialysis
* Child C cirrhosis of the liver
* Known genetic cardiomyopathies

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study Population: Peri and postmenopausal women with cardiovascular disease or high risk for CVD with and without hormon replacement therapy
Study Population: Study Population: Peri and postmenopausal women with cardiovascular disease or high risk for CVD with and without hormon replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 2725 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2035-03 (Estimated); Study Completion 2035-03 (Estimated)

PRIMARY OUTCOMES:
MACCE | 10 years
  defined as death, cardiovascular death, myocardial infarction, stroke, Transient Ischemic Attack, revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, MD, Study Director — Division of Cardiology, Pulmonary Disease and Vascular Medicine at University Hospital Duesseldorf; Lisa Dannenberg, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine at University Hospital Duesseldorf
Locations (2):
- Germany (2):
  - Clinic for Cardiology, Angiology and Intensive Care at Charité Mitte Berlin, Berlin
  - University Hospital Duesseldorf, Düsseldorf

IPD SHARING:
Plan to Share IPD: No
not necessary